CLINICAL TRIAL: NCT06849648
Title: The Effect of Buzzy and Finger Puppet Show on Children's Pain, Fear, and Anxiety During Venipuncture in the Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: Impact of Buzzy and Finger Puppets on Children's Pain, Fear, and Anxiety During Venipuncture
Acronym: Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Mardin Artuklu University (Other); Bartın Unıversity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0000000000000000000002024/11-3
Record Dates: First submitted 2025-01-24; First posted 2025-02-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Pain Management; Nonpharmalogical Pain Management; Children Pain Management
Keywords: Buzzy device; finger puppets; nonpharmacologic methods; pain management in children; Pediatric venipuncture
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This study used a parallel, randomized, double-blind design to evaluate the effects of the Buzzy device and finger puppets on pain, fear, and anxiety in children aged 4-7 undergoing venipuncture.
  Participants were randomly assigned to the Buzzy Group (Buzzy device applied during venipuncture), Puppet Group (distraction with finger puppets), or Control Group (no intervention).
  Standardized venipuncture procedures were performed by an experienced pediatric nurse. Pain, fear, and anxiety levels were assessed before and one minute after the procedure using child-friendly scales (Wong-Baker Faces Pain Scale, Children's Fear Scale, and Children's Anxiety Meter-State (CAM-S)).
Who Masked: Participant, Investigator
Masking Description: Participant: The participant doesn't know their group assignment.
  Investigator: The researcher analyzing the data or designing the study is blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental A (Experimental): the Buzzy device, shaped like a bee or ladybug and featuring a reusable battery, was used for pain management. The device combines cold application with vibration, aided by wing-shaped ice packs. We used the ladybug-shaped Buzzy (Buzzy Healthcare mini ladybuzz, code BKHM3). Following the manufacturer's instructions, the device was held 3-5 cm above the venipuncture site for 30 seconds, then moved just before injection while maintaining vibration throughout the procedure. Ice packs were kept in the freezer but were removed a few minutes before the procedure to avoid discomfort from excessive cold. After the procedure, the device was cleaned with alcohol, and the ice pack was placed back in the freezer for reuse. The total intervention lasted 2-5 minutes, with parents present but not allowed to soothe their children during the procedure.
  Interventions: Device: The Buzzy Device
- Experimental B (Experimental): Finger puppets were used to distract the participants during venepuncture procedure. Children are allowed to pick their favourite animals. These soft in various shaped finger puppets can be placed on adult's fingers. One minute before the venipuncture procedure, the researcher (K.O.) engaged the participants in finger puppet play and initiated conversation by asking; 'Hello, how are you? What is this figure? Do you know where this animal/figure live in? Have you previously seen this animal/figure alive? Have you been in a zoo? Additionally, techniques such as having the animals 'sing' or 'interact' with each other were employed to capture the child's attention on the finger puppets. Children in this group were not given any distraction techniques prior to the procedure. All groups' parents accompanied over their children during the process, but they were not permitted to comfort them.
  Interventions: Device: Finger Puppet
- Control Group: No intervention is applied; participants receive the standard venipuncture procedure. (No Intervention): Children in this group were invited for venipuncture procedure in accordance with the standard venipuncture procedure applied in the paediatric emergency department and the procedure was performed. Similarly to intervention groups, any distraction did not used, or families were not allowed to comfort their children during procedure. In this scale, faces are given a pain score according to numerical values.

INTERVENTIONS:
Device: The Buzzy Device — In essence, the Buzzy device offers a multi-sensory approach (vibration + cold) in conjunction with a hygienic protocol, which is a key differentiator from other non-pharmacological interventions such as distraction through toys, videos, or verbal techniques. Currently, there is no studies evaluating the use of the Buzzy device and finger puppets, which are nonpharmacologic methods, in relation to the levels of pain, fear, and anxiety in children aged 4-7 years undergoing venipuncture procedures in emergency department settings.
  Arms: Experimental A
Device: Finger Puppet — Finger puppets were used to distract the participants during venepuncture procedure. Children are allowed to pick their favourite animals. These soft in various shaped finger puppets can be placed on adult's fingers. One minute before the venipuncture procedure, the researcher (K.O.) engaged the participants in finger puppet play and initiated conversation by asking; 'Hello, how are you? What is this figure? Do you know where this animal/figure live in? Have you previously seen this animal/figure alive? Have you been in a zoo? Additionally, techniques such as having the animals 'sing' or 'interact' with each other were employed to capture the child's attention on the finger puppets. Children in this group were not given any distraction techniques prior to the procedure. All groups' parents accompanied over their children during the process, but they were not permitted to comfort them.
  Arms: Experimental B

SUMMARY:
This study evaluates the impact of the Buzzy device and finger puppet distraction on pain, fear, and anxiety in children aged 4-7 undergoing venipuncture in a pediatric emergency department. Designed as a parallel, randomized, double-blind clinical trial, participants were divided into three groups: Buzzy Group (BG), Puppet Group (PG), and a Control Group (CG).

The Buzzy Group used the Buzzy device during venipuncture, the Puppet Group received finger puppet distraction, and the Control Group underwent standard venipuncture with no intervention. Pain, fear, and anxiety levels were assessed before and one minute after venipuncture using child-friendly scales, including the Wong-Baker Faces Pain Scale, Children's Fear Scale (CFS), and Children's Anxiety Meter-State (CAM-S).

All procedures were performed by an experienced pediatric nurse trained in Buzzy device usage. Recruitment took place at Mardin Training and Research Hospital from January to June 2025, focusing on children aged 4-7 without chronic illnesses, neurodevelopmental delays, or other exclusion criteria such as prior sedation or cold sensitivity disorders. Parents and children in the intervention groups were educated about the respective techniques in age-appropriate language.

This trial aims to compare the effectiveness of these nonpharmacologic interventions in reducing procedural distress, providing evidence-based solutions for managing pain and anxiety in pediatric emergency settings.

DETAILED DESCRIPTION:
This study investigates the effectiveness of the Buzzy device and finger puppets-nonpharmacologic methods-in reducing pain, fear, and anxiety in children aged 4-7 undergoing venipuncture in emergency departments, addressing a gap in current research.

This study was designed as a parallel, randomized and double-blind clinical trial on pediatric patients. Patients who needed to undergo a venipuncture procedure by the emergency nurse were randomly assigned to three different groups: Intervention Group 1 (use of Buzzy device, referred to as Buzzy Group [BG]), Intervention Group 2 (distraction with a finger puppet, referred to as Puppet Group [PG]), and the Control Group referred to as [CG].

Patients in Intervention Group 1 received the Buzzy device during venipuncture, while patients in Intervention Group 2 received distraction with finger puppets. Patients in the Control Group did not receive any intervention. Patients in all groups were subjected to the standard venipuncture procedure.

Children's pain, fear and anxiety levels were assessed by using Wong-Baker Faces Pain Rating Scale, Children's Fear Scale (CFS), Children's Anxiety Meter-State (CAM-S) before and 1 minutes after the venipuncture procedure. These assessments were performed independently by the children themselves.

All venipuncture procedures were carried out by the same nurse who are working in the paediatric emergency ward and had at least eight years of experience with the paediatric venipuncture procedure. Additionally, the nurse received training on how to operate the Buzzy device during venipuncture procedure. Venipuncture was performed with the peripheral venous line.

This method aims to compare the effect of different distraction techniques on children's pain and anxiety levels during venipuncture.

The children were recruited from the paediatric emergency departments of Mardin Training and Research Hospital, in the city of Mardin, in the Southeastern Anatolia Region of Turkey, between January 2025 and June 2025.

In this study, we included samples of patients aged 4-7 years of both genders who had been admitted to the paediatric emergency ward. These children required venepuncture procedures for blood tests. The study excluded the children who with chronic disease; who were neuro-developmentally delayed verbal difficulties, hearing or visual impairments; children who had received analgesia or sedation within the previous 24 hours, or had a history of syncope and those were unconscious. Also, children who have bleeding disorder; and infection, rash, damaged skin on the arm where the device will be placed will be excluded from the study. In addition, children with cold sensitivity disease such as Raynaud's disease and Prader-Willi syndrome and children who refuse to wear the Buzzy device were excluded from the study.

The researcher evaluated participants' baseline information in order to analyse eligibility requirements. Parents of participants in the intervention 1. and 2. groups were informed that Buzzy device and finger puppet play, respectively, would be used for their kids during venipuncture, respectively. Additionally, the participants were informed how to use the Buzzy device and finger puppet play during venipuncture with an age-appropriate language. In the control group, parents were informed that only children's pain, fear and anxiety would be measured before and after the venipuncture procedure. To prevent measurement bias, no additional information was provided to the nurses, the participants and their families.

ELIGIBILITY:
Inclusion criteria:

* In this study, we included samples of patients aged 4-7 years of both genders who had been admitted to the paediatric emergency ward.
* These children required venepuncture procedures for blood tests.

Exclusion criteria:

* The study excluded the children who with chronic disease; who were neuro-developmentally delayed verbal difficulties, hearing or visual impairments;
* Children who had received analgesia or sedation within the previous 24 hours, or had a history of syncope and those were unconscious.
* Children who have bleeding disorder; and infection, rash, damaged skin on the arm where the device will be placed will be excluded from the study.
* Children with cold sensitivity disease such as raynaud's disease and prader-willi syndrome and children who refuse to wear the buzzy device were excluded from the study.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
The Best Pain Management Method | up to 5 months
  Pain Level: Measured using the Wong-Baker Faces Pain Rating Scale and Visual
  This numerical rating scale spans from 0 to 5, with facial expressions representing emotions ranging from a smiling face (0 = very happy/no pain) to a crying face (5 = worst pain)

SECONDARY OUTCOMES:
Fear Metrics: Understanding and Measuring the Emotion | up to 5 months
  Fear Level: Assessed using the Children's Fear Scale (CFS), which is designed to gauge a child's level of fear before and after the procedure.
  Face 0 'no scared at all'; Face 1 'a little bit more scared'; Face 2 'a bit more scared'; Face 3 'more scared', Face 4 'severe scared' (Figure 3).Therefore, scale scoring ranges from neutral (0=no scared) to frightened (4=severe scared), indicating that as the score increases, the level of fear increases.

OTHER OUTCOMES:
Anxiety Assessment in Children: Using the CAM-S for Pre- and Post-Procedure Evaluation | up to 5 months
  Anxiety Level: Measured by the Children's Anxiety Meter-State (CAM-S), which evaluates the anxiety levels of the child before and 1 minute after the procedure.
  Scores range from 0 to 10, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: AHMET BUTUN, PhD, Principal Investigator — Mardin Artuklu University
Locations (1):
- Mardin Training and Research Hospital, Mardin, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing IPD could potentially breach participant confidentiality, especially if sensitive personal data is involved. Ethical guidelines and data protection regulations (e.g., GDPR) require that personal data be kept confidential.

REFERENCES:
- See also: Nonpharmacological pain management uses techniques to reduce pain and anxiety without medications. This guide covers common strategies for children, the role of parents as coaches, age-specific methods, and considerations for chronic pain and development — https://pmc.ncbi.nlm.nih.gov/articles/PMC6179554/